CLINICAL TRIAL: NCT07303140
Title: Non-invasive Assessment of Liver Fibrosis in a French Cohort of Pediatric Patients With Type III Glycogen Storage Disease: Current State and Perspectives
Acronym: HEPAGLY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9479
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Liver Fibrosis
Keywords: Liver fibrosis; Type III glycogen storage disease; Liver fibrosis in pediatric patients
MeSH Terms: conditions — Liver Cirrhosis; Glycogen Storage Disease Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with type III glycogen storage disease (GSDIII) can develop liver fibrosis, which can be complicated by liver failure or even hepatocellular carcinoma. Since the beginning of the 21st century, non-invasive techniques for assessing fibrosis, such as liver elastography, have been developed. These techniques often make it possible to avoid liver biopsies during patient follow-up and have already been validated in the management of several diseases in adults. These techniques are also beginning to be recommended for monitoring certain chronic liver diseases in children.

ELIGIBILITY:
Inclusion Criteria:

* Minors: from birth to 17 years
* Adults: 18 to 21 years
* Subjects being monitored for type III glycogen storage disease and having had at least one liver elastography measurement during their follow-up.

Exclusion Criteria:

- Patients monitored for type III glycogen storage disease but who had never undergone liver elastography during their follow-up.

Ages: 1 Month to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients under 22 years of age
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Liver elastography values | 1 hour after consultation
  Liver fibrosis is classified into four stages, from 0 to 4:
  * F0 corresponds to the absence of fibrosis
  * F4 corresponds to established cirrhosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France